CLINICAL TRIAL: NCT01976065
Title: Regeneration of Pulp-Dentin Development in Teeth With Necrotic Pulps and Immature Roots
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kenneth Hargreaves (Other)
Collaborators: University of Maryland, Baltimore (Other); Loma Linda University (Other); University of North Carolina (Other); American Association of Endodontists (Other)
Responsible Party: Sponsor-Investigator, Kenneth Hargreaves, Chair, Dept. of Endodontics, UTHSCSA, The University of Texas Health Science Center at San Antonio
Organization: The University of Texas Health Science Center at San Antonio (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: HSC20130467H
Record Dates: First submitted 2013-10-29; First posted 2013-11-05 (Estimated); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Pulp Necrosis; Regeneration
Keywords: Necrotic tooth pulp; Immature permanent teeth; Regeneration
MeSH Terms: conditions — Dental Pulp Necrosis | interventions — Ciprofloxacin; Metronidazole; Minocycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Mineral Trioxide Aggregate (MTA) (Other): Standard Treatment group consisting of placement of Mineral Trioxide Aggregate (MTA), an FDA approved dental material at the end of an immature root followed by a composite restoration (crown).
  Interventions: Other: Standard Treatment
- Revascularization Treatment (REVASC) (Experimental): Consists of standard treatment procedure PLUS disinfection of the canal space with Triple Antibiotic Paste study medication followed by placement of Collaplug, an FDA approved material to help promote clotting. A composite restoration in then placed.
  Interventions: Drug: Triple Antibiotic Paste
- Regeneration Treatment (REGENDO) (Experimental): Consists of standard treatment procedure PLUS Triple Antibiotic Paste study medication PLUS use of Emdogain, an FDA approved medication used in an FDA approved manner, that is a growth factor to help surrounding tissues to grow together and heal.
  Interventions: Drug: Triple Antibiotic Paste

INTERVENTIONS:
Drug: Triple Antibiotic Paste — USP antibiotic drugs mixed at a 1:1:1 ratio into a powder that is mixed with sterile saline to a paste-like consistency
  Other Names: Ciprofloxacin, Metronidazole, & Minocycline
  Arms: Regeneration Treatment (REGENDO); Revascularization Treatment (REVASC)
Other: Standard Treatment — Standard Treatment no use of study drug
  Other Names: No use of study drug
  Arms: Mineral Trioxide Aggregate (MTA)

SUMMARY:
This multi-center exploratory clinical trial is a randomized trial designed to test whether a regenerative endodontic procedure using tissue engineering principles (REGENDO), or a revascularization (REVASC) endodontic procedure, in comparison to standard apexification treatment using a mineral trioxide aggregate barrier (apexification; APEX), produces a significantly better composite clinical outcome for the treatment of immature permanent teeth with pulpal necrosis.

DETAILED DESCRIPTION:
This is a multi-center randomized clinical trial designed to test whether a regenerative endodontic procedure using tissue engineering principles (REGENDO), or a revascularization (REVASC) endodontic procedure, when compared to the standard apexification treatment using mineral trioxide aggregate barrier-MTA apexification (APEX), produces a significantly better composite clinical outcome for the treatment of immature permanent teeth with pulpal necrosis. This study will use an antibiotic mixture called Triple Antibiotic Paste (TAP), consisting of ciprofloxacin, metronidazole and minocycline, in the tooth for disinfection of the root canal in study arms REGENDO and REVASC. The FDA has issued an Investigational New Drug (IND) number allowing use of the triple antibiotic mixture in this trial. Other dental materials used in this study have already been FDA approved for use in humans to provide a matrix for the promotion of tissue growth in the root canal space. The study will also attempt to identify the type of bacteria within the root canal space and surrounding tissues by analyzing a small sample collected on a cotton-tip applicator. This clinical trial hopes to determine which of the three treatment methods helps the tooth to grow stronger and survive for at least two years after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-20
* Participant has a permanent tooth with a necrotic pulp (as defined by lack of responsiveness to both electrical pulp tests and cold [EndoIce] tests). If the tooth was traumatized, then pulpal necrosis is defined as either: 1) no response to both electrical pulp test and cold [EndoIce] test by three months after trauma, or 2) presence of a periapical lesion, or 3) radiographic evidence of root resorption, or 4) discoloration of the crown.
* Tooth in question is restorable (as defined by Class A or Class B using Samet and Jotkowitz classification) without the need of a stainless steel crown.
* Incomplete (i.e., immature) root development defined by apical foramen ≥1.0mm (each foramina >1.0mm for multi-rooted teeth).
* At least 5 mm of root development (CEJ to radiographic apex).
* Willing and able to provide informed assent/consent.
* Legal guardian willing and able to provide informed consent.

Exclusion Criteria:

* No access to telephone for study contacts.
* Unable to comprehend study materials in English or Spanish.
* Subject not available for follow up at 12 or 24 months.
* Previous allergic response to ciprofloxacin, metronidazole or minocycline or any materials used in the study.
* History of systemic diseases with altered immune function including diabetes, immunodeficiency, leukemia, Addison's or Cushing's disease.
* History of taking immunosuppressants or chemotherapeutic agents including glucocorticoids in the past 3 months.
* Clinical or radiographic evidence of root fracture or alveolar fracture.
* Tooth in question received prior endodontic obturation.
* Tooth in question has class III mobility or dens invaginatus.
* Tooth in question has a history of avulsion with extra-oral dry time longer than 1 hour.
* Clinical judgement (with documentation of the reason)
* Radiographic or clinical identification of ankylosis (replacement resorption) or inflammatory (infection-related) root resorption.

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 125 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2018-09-24 (Actual); Study Completion 2018-09-24 (Actual)

PRIMARY OUTCOMES:
Tooth Survival | 2 years
  1) the growth in hard tissue deposition in the radiographic root area is increased by at least 20%, and 2) the tooth survives to this time point and 3) there is no pain.

SECONDARY OUTCOMES:
Positive pulpal response | 2 years
  Comparison of treatment effects on positive pulpal responses, crown staining, preoperative factors (age, sex, history of trauma), or antimicrobial efficacy and residual intracanal microbial load would influence the primary outcome measure of tooth survival.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Hargreaves, DDS, PhD, Study Chair — University of Texas
Locations (4):
- United States (4):
  - Loma Linda University, Loma Linda, California
  - University of Maryland, Baltimore, Maryland
  - University of North Carolina, Chapel Hill, North Carolina
  - University of Texas Health Science Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
No plan to share data at this time.